CLINICAL TRIAL: NCT03333694
Title: A Randomized Investigator and Patient Blind Placebo-controlled Parallel Group First in Human and Proof of Concept Study to Evaluate the Safety Tolerability and Efficacy of CLL442 in Patients With Cutaneous Squamous Cell Carcinoma in Situ
Brief Title: Safety, Tolerability, and Efficacy Study of CLL442 in Patients With Cutaneous Squamous Cell Carcinoma in Situ (SCCis)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study fully enrolled and completed after last patient completed the study
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCLL442X2201
Record Dates: First submitted 2017-10-12; First posted 2017-11-07 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-09

CONDITIONS: Cutaneous Squamous Cell Carcinoma in Situ (CSCCis)
Keywords: Cutaneous Squamous Cell Carcinoma (cSCC) in situ, mTOR kinase inhibitors, PI3K inhibitor.

STUDY DESIGN:
Intervention Model Description: A first in human,proof of concept study. The study is investigator-and patient-blinded, randomized, placebo-controlled study in patients with SCCis, to assess safety, tolerability and initial efficacy of CLL442 after up to 84 days twice daily application of CLL442 or placebo on one lesion.
Who Masked: Participant, Investigator
Masking Description: investigator and patient blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLL442 (Experimental): Cutaneous Cream application twice daily
  Interventions: Drug: Cutaneous Cream application
- Placebo (Placebo Comparator): Placebo Cutaneous Cream application twice daily
  Interventions: Drug: Placebo Cutaneous Cream application

INTERVENTIONS:
Drug: Cutaneous Cream application — Cutaneous Cream application twice daily with experimental (CLL442)
  Arms: CLL442
Drug: Placebo Cutaneous Cream application — Cutaneous Cream application twice daily with placebo
  Arms: Placebo

SUMMARY:
The purpose of this first in human and proof of concept study is to characterize the safety, tolerability and initial efficacy of CLL442 in patients with Squamous Cell Carcinoma in situ (SCCis) to enable further clinical development of CLL442.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained.
2. Male and female patients, age ≥ 18 to ≤ 90 years (at the time of the screening visit).
3. A primary, clinically diagnosed and histologically confirmed cutaneous SCC in situ lesion, with or without the involvement of the follicular unit, and histologically diagnosed within 30 days of the screening visit. The post-biopsy residual SCCis lesion must be visually evident and at least 3 mm in either length or width.
4. The lesion must be located in a place easily accessible for topical application by the patient or their caregiver, excluding the genitals, perianal area, sub-ungual area, eyelids, ear and must be >1 cm away from the eyes and mouth.

Exclusion Criteria:

1. Evidence of dermatological disease or histological evidence of a confounding skin condition in the treatment area, including but not limited to BCC, worse level/grade of SCC, rosacea, psoriasis, atopic dermatitis, eczema, xeroderma pigmentosa, verrucous lesions or any other tumor in the biopsy specimen. Lesions with atypical histology such as: spindle cell SCC, acantholytic SCC, clear cell SCC, adenosquamous SCC, desmoplastic SCC or lesions that have been present for a short time and have been fast growing.
2. Treatment of the target SCCis lesion within 8 weeks of screening visit by any of the following treatments: Liquid nitrogen, Photochemotherapy (PUVA), Long wave ultra violet radiation (UVB light), surgical excision or curettage within 1 cm of target lesion.; Systemic retinoids.; Ionizing radiation or interlesional injections or; Undergone a facial resurfacing procedure, i.e., chemical peel, laser resurfacing, dermabrasion, within the target lesion;
3. Treatment with the following topical agents within the 4 weeks prior to the screening visit: Levulanic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, hyaluronic acid, imiquimod.
4. History of recurrence of the target SCCis lesion.
5. Systemic use of immunosuppressive drugs within 4 weeks prior to screening visit or during the treatment period - Photodynamic therapy or immunomodulators, cytotoxic drugs, or interferon/interferon inducers within 4 weeks prior to study entry or expected during the study.
6. Women of child-bearing potential, unless they are using at least basic methods of contraception during dosing of investigational drug.
7. Pregnant or nursing (lactating) women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE), serious adverse events (SAEs) of CLL442 on lesion free skin at Day 7 | Day 7
  As part of safety and tolerability assessment, assess the incidence of adverse events (AE), serious adverse events (SAEs) in patients with SCCis treated with CLL442 or placebo on lesion free skin for 7 days
Change in the size of One SCCis lesion area at Day 84 from Day 1 | Day 1 and Day 84
  Area is measured by pen and ruler and standardized digital photography
Change in the Local skin reactions severity score at Day 7 or Day 84 from Day 1 | Day 1, Day 7, Day 84
  Local skin reactions severity score
Incidence of adverse events (AE), serious adverse events (SAEs) of CLL442 on SCCis lesion at Day 84 | Day 84
  As part of safety and tolerability assessment, assess the incidence of adverse events (AE), serious adverse events (SAEs) in patients with SCCis treated with CLL442 or placebo on SCCis lesion area for 84 days.

SECONDARY OUTCOMES:
CLL442 plasma concentration | Day 1 through Day 84
  To evaluate the systemic pharmacokinetics of CLL442
Time required to achieve 50% decrease in 1 lesion area. | 84 days
  Part of efficacy assessment.
Time required to achieve complete SCCis 1 lesion clearance (censored by end of study visit). | 84 days
  Part of efficacy assessment.
Percentage of pts with complete clearance at the end of the study, assessed visually and histologically | 84 days
  Part of efficacy assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (3):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Gainesville, Florida
- Australia (3):
  - Novartis Investigative Site, Phillip, Australian Capital Territory
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Benowa, Queensland
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CCLL442X2201 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17537
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=482